CLINICAL TRIAL: NCT02393937
Title: A Multi-center, Double-blind, Randomized, Vehicle-controlled, Parallel-group Study Comparing Metronidazole Gel 1%, to Metrogel® (Metronidazole Gel) 1% in the Treatment of Rosacea
Brief Title: A Therapeutic Equivalence Study of Two Metronidazole Gel 1% Topical Treatments of Rosacea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: bioRASI, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LO-17-3-2014
Record Dates: First submitted 2015-03-12; First posted 2015-03-20 (Estimated); Last update posted 2020-09-03 (Actual); Status verified 2016-11

CONDITIONS: Papulopustular Rosacea; Erythematotelangiectatic Rosacea
MeSH Terms: conditions — Rosacea | interventions — Metronidazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Test: Metronidazole Gel 1% (Experimental): Metronidazole Gel 1% once daily for 70 days.
  Interventions: Drug: Test: Metronidazole Gel 1%
- Reference: Metronidazole Gel 1% (Active Comparator): Metronidazole Gel, 1% (MetroGel) Galderma S.A. once daily for 70 days.
  Interventions: Drug: Reference: Metronidazole Gel 1%
- Placebo (Placebo Comparator): Placebo Gel once daily for 70 days.
  Interventions: Drug: Placebo Gel

INTERVENTIONS:
Drug: Reference: Metronidazole Gel 1% — Participants are assigned to one of three groups in parallel for the duration of the study
  Other Names: MetroGel
  Arms: Reference: Metronidazole Gel 1%
Drug: Test: Metronidazole Gel 1% — Participants are assigned to one of three groups in parallel for the duration of the study
  Arms: Test: Metronidazole Gel 1%
Drug: Placebo Gel — Participants are assigned to one of three groups in parallel for the duration of the study
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare the efficacy of two Metronidazole Gels 1%, in the treatment of Rosacea.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female subjects with at least 18 years of age;
* Read and signed ICF;
* Clinical Diagnosis of Rosacea;

Exclusion Criteria:

* Females who are pregnant, lactating or of childbearing potential who are not using or do not agree to use an acceptable form of contraception;
* Any skin condition that would interfere with treatment of rosacea
* Use of prohibited medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 963 (Actual)
Dates: Start 2015-02; Primary Completion 2015-07 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
To compare the test and reference products of metronidazole topical gel 1% with regard to the mean percent change from Baseline of the inflammatory lesion counts of rosacea. | 70 Days

SECONDARY OUTCOMES:
To compare the test and reference product of metronidazole topical gel 1% with regard to the Investigator's Global Evaluation (IGE) of disease severity | 70 Days

CONTACTS AND LOCATIONS:
Locations (26):
- United States (26):
  - Los Angeles, California
  - San Diego, California
  - Boca Raton, Florida
  - Clearwater, Florida
  - Miami, Florida
  - Miramar, Florida
  - Ocala, Florida
  - Tampa, Florida
  - Lexington, Kentucky
  - Watertown, Massachusetts
  - Las Vegas, Nevada
  - New York, New York
  - High Point, North Carolina
  - Raleigh, North Carolina
  - Cincinnati, Ohio
  - Philadelphia, Pennsylvania
  - Warwick, Rhode Island
  - Mt. Pleasant, South Carolina
  - Austin, Texas
  - El Paso, Texas
  - Houston, Texas
  - Pflugerville, Texas
  - Plano, Texas
  - San Antonio, Texas
  - Arlington, Virginia
  - Norfolk, Virginia